CLINICAL TRIAL: NCT05015322
Title: Comparison of the Effectiveness of the Ultrasound Guided Subacromial, Acromioclavicular With Subacromial Injection and Suprascapular Nerve Block in Patients With Shoulder Impingement Syndrome ; A Randomized Controlled, Single Blind, Clinical Trial
Brief Title: Comparison of the Effectiveness of the Ultrasound Guided Injections in Patients With Shoulder Impingement Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Burcu Metin Ökmen, Principal Investigator,Assoc.Phd.M.D., Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BYIEAH2
Record Dates: First submitted 2021-08-18; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Shoulder Impingement; Ultrasound Guided Injection
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Bupivacaine; Methylprednisolone

STUDY DESIGN:
Intervention Model Description: prospective,randomized controlled, single blind
Who Masked: Outcomes Assessor
Masking Description: The patients were followed up and questioned by the evaluator, who was blind to the type of injection administered to the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- subacromial injection (Active Comparator): ultrasound (US)-guided subacromial injection
  Interventions: Drug: bupivacaine and methylprednisolone
- acromioclavicular joint and subacromial injection (Active Comparator): ultrasound (US)-guided acromioclavicular joint and subacromial injection
  Interventions: Drug: bupivacaine and methylprednisolone
- suprascapular nerve block (Active Comparator): ultrasound (US)-guided suprascapular nerve block
  Interventions: Drug: bupivacaine and methylprednisolone

INTERVENTIONS:
Drug: bupivacaine and methylprednisolone — 5 mL of 0.25% bupivacaine containing 20 mg methylprednisolone was administered to the subacromial area
  Arms: subacromial injection
Drug: bupivacaine and methylprednisolone — 5 mL of 0.25% bupivacaine containing 20 mg methylprednisolone was administered to the subacromial area for the subacromial+acromioclavicular joint injection. In addition, 2 mL of 20 mg methylprednisolone and the same concentration of local anaesthetic were injected into the acromioclavicular joint
  Arms: acromioclavicular joint and subacromial injection
Drug: bupivacaine and methylprednisolone — suprascapular nerve block was administered with a mixture of 10 mL of 0.25% bupivacaine and 40 mg methylprednisolone
  Other Names: suprascapular nerve block
  Arms: suprascapular nerve block

SUMMARY:
Shoulder pain, which is the third most common cause of musculoskeletal pain, has different etiologies. Muscle, bone structures and connective tissue pathologies can cause shoulder pain. Impingement syndrome (IS), which can cover many terms such as rotator cuff disorders, tendinitis and tears, is one of the most common pathologies of shoulder pain.

DETAILED DESCRIPTION:
The hypothesis of this study was that injection types including ACJ would increase treatment efficacy.Therefore, this study investigated the six-month follow-up results of patients undergoing SA injection and SSNB and those receiving SA and ACJ injection.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-65,
* who were suffering from shoulder pain for more than three months and
* who were diagnosed with IS.
* All patients included in the study were diagnosed with IS using Shoulder Magnetic Resonance imaging.

Exclusion Criteria:

* the presence of cervical radiculopathy;
* undergoing shoulder operation before;
* the presence of central nervous system or
* the presence of rheumatological disease, and polyneuropathy;
* receiving physical therapy in the shoulder area with a diagnosis of IS within the last six months; and
* receiving any injection therapy in the past.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | six month
  for pain. 0: no pain at all, 10: worst pain imaginable

SECONDARY OUTCOMES:
Shoulder pain and disability index (SPADI) | six month
  This scale was developed to measure pain and disability associated with shoulder pain. It consists of two parts evaluating pain and disability.
Short-Form 12 (SF-12) | six month
  The SF-12 has a physical (SF12-PCS) and mental (SF12-MCS) state assessment scale

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Metin Ökmen, Assoc. Prof, Principal Investigator — University of Health Sciences, Yuksek Ihtisas Training and Research Hospital; Korgün M Ökmen, Assoc. Prof, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital